CLINICAL TRIAL: NCT02458781
Title: Antibiotic Treatment Trial for Small Intestinal Bacterial Overgrowth: A Randomized, Double-Blind, Placebo-Controlled Trial Comparing Ciprofloxacin and Metronidazole
Brief Title: Antibiotic Treatment Trial for Small Intestinal Bacterial Overgrowth
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: San Antonio Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Karin S. Gilkison, Gastroenterology Fellow, San Antonio Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 398092-1
Record Dates: First submitted 2015-04-10; First posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Small Intestinal Bacterial Overgrowth
MeSH Terms: interventions — Metronidazole; Ciprofloxacin; Fluoroquinolones; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo capsule:
  To be provided by BAMC Pharmacy. It will be made and stored by BAMC pharmacy. The matching placebo will be a gelatin capsule filled with methylcellulose powder only. Patient will take 2 capsules two times a day for 14 days.
  Interventions: Drug: Placebo
- Ciprofloxacin (Active Comparator): Ciprofloxacin 250mg capsule:
  To be provided by BAMC pharmacy. It will be made and stored by BAMC Pharmacy. Ciprofloxacin 250mg tablet will be encapsulated with a gelatin capsule filled with methylcellulose. Patient will take 2 capsules of Ciprofloxacin 250mg two times a day for 14 days.
  Interventions: Drug: Ciprofloxacin
- Metronidazole (Active Comparator): Metronidazole 250mg capsule:
  To be provided by BAMC pharmacy. It will be made and stored by BAMC Pharmacy. Metronidazole 250mg will be encapsulated with a gelatin capsule filled with methylcellulose. Patient will take 2 capsules of metronidazole 250mg two times a day for 14 days.
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Metronidazole — Metronidazole 500mg given twice daily for 14 days
  Other Names: flagyl; metro
  Arms: Metronidazole
Drug: Ciprofloxacin — Ciprofloxacin 500mg given twice daily for 14 days
  Other Names: cipro; fluoroquinolone
  Arms: Ciprofloxacin
Drug: Placebo — Placebo given twice daily for 14 days
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to evaluate the efficacy of ciprofloxacin versus metronidazole versus placebo in eradication of small intestinal bacterial overgrowth (SIBO).

DETAILED DESCRIPTION:
Approximately 180 study subjects with SIBO identified by positive glucose hydrogen breath (GHB) testing who meet inclusive and exclusive criteria will be randomized to receive either ciprofloxacin 500mg by mouth twice daily, metronidazole 500mg by mouth twice daily, or placebo by mouth twice daily. Subjects will complete a baseline symptom questionnaire and be treated for 14 days. Response will be assessed at end of treatment. The Gastrointestinal Symptom Rating Scale (GSRS) and GHB testing will be performed at the end of treatment. Subjects with a negative GHB at the end of treatment are considered as cured, or treatment success. Patients with treatment success will be reassessed for long-term response to treatment or disease recurrence at 30 days, 4 months, and 9 months using GHB. Symptoms will also be re-assessed at the 30 day, 4 month, and 9 month intervals with GSRS-IBS symptom questionnaire done prior to GHB testing.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age greater than 18 who have been diagnosed with SIBO after a clinically indicated hydrogen breath test.
* Patients with liver disease or liver cirrhosis will be included, as this particular group is at higher risk for developing SIBO, would potentially benefit from inclusion, and do not require dose adjustments with either study medication.
* Patients on warfarin are not excluded, but INR will be uniformly recommended to be checked within 1 week of therapy initiation, as standard practice through the Coumadin clinic, for the potential effect on INR and increased risk of bleeding while on any antibiotic

Exclusion Criteria:

* Patient age less than 18
* Hypersensitivity to the antibiotics
* Pregnancy or breast feeding
* Patients who cannot consent for themselves
* End stage renal disease defined as creatinine clearance <30 mL/min or on hemodialysis.
* Patients who have taken antibiotics in the past 30 days
* Laxatives, stool softeners, or bulk fiber in the last 7 days
* Enemas or suppositories in the last 3 daysⱡ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients cured of SIBO after treatment with ciprofloxacin versus metronidazole versus placebo. | 2 weeks

SECONDARY OUTCOMES:
Gastrointestinal symptoms based on questionnaire | Immediately post-treatment (approximately 2 weeks), 30 days, 4 months, and 9 months
Disease relapse rate of SIBO after treatment success | Immediately post-treatment (approximately 2 weeks), 30 days, 4 months, and 9 months
Time interval between treatment success and recurrence of SIBO | Immediately post-treatment (approximately 2 weeks), 30 days, 4 months, and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Karin S Gilkison, MD, MPH, Principal Investigator — Gastroenterology Fellow